CLINICAL TRIAL: NCT01153841
Title: Primary Vaccination Course With the Pneumococcal Vaccine GSK 1024850A, in Healthy Infants in Vietnam When Co-administered With GSK Biologicals' Infanrix Hexa™ (DTPa-HBV-IPV/Hib) Vaccine
Brief Title: Primary Vaccination Study With GSK Biologicals' Pneumococcal Vaccine in Healthy Infants in Vietnam
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 113151; 2012-000162-38 (EudraCT Number)
Record Dates: First submitted 2010-06-17; First posted 2010-06-30 (Estimated); Results first posted 2017-02-27 (Actual); Last update posted 2020-01-02 (Actual); Status verified 2019-12

CONDITIONS: Infections, Streptococcal; Streptococcus Pneumoniae Vaccines
Keywords: Pneumococcal vaccine
MeSH Terms: conditions — Streptococcal Infections | interventions — diphtheria-tetanus-acellular pertussis-inactivated poliovirus-Haemophilus influenzae b conjugate-hepatitis B vaccine

ARMS (2):
- Synflorix Group (Experimental): Subjects receiving Synflorix™(GSK 1024850A) co-administered along with Infanrix hexa™.
  Interventions: Biological: Synflorix™( GSK1024850A); Biological: Infanrix hexa™
- Control Group (Active Comparator): Subjects receiving Infanrix hexa™ vaccine alone.
  Interventions: Biological: Infanrix hexa™

INTERVENTIONS:
Biological: Synflorix™( GSK1024850A) — Intramuscular, 3 doses
  Arms: Synflorix Group
Biological: Infanrix hexa™ — Intramuscular, 3 doses

SUMMARY:
The purpose of the study is to evaluate the safety and reactogenicity of Synflorix™ (GSK 1024850A) given as a 3-dose primary immunization course when co-administered with Infanrix hexa™ vaccine at 2, 3 and 4 months of age in infants in Vietnam.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subjects between, and including 6-12 weeks of age at the time of the first vaccination.
* Subjects for whom the investigator believes that their parents/guardians can and will comply with the requirements of the protocol.
* Written and signed or thumb-printed informed consent obtained from the parent(s)/LAR of the child. Where parent(s)/guardian(s) are illiterate, the consent form will be countersigned by a witness.
* Free of obvious health problems as established by medical history and clinical examination before entering into the study.

Exclusion Criteria:

* Use of any investigational or non-registered product other than the study vaccine(s) within 30 days preceding the first dose of study vaccine, or planned use during the study period.
* Concurrently participating in another clinical study, at any time during the study period, in which the subject has been or will be exposed to an investigational or a non-investigational product.
* Acute disease and/or fever at the time of enrolment.
* History of any reaction or hypersensitivity likely to be exacerbated by any component of the vaccine(s).
* History of chronic condition(s) requiring treatment such as cancer or autoimmune disease.
* Hypersensitivity to latex.
* Previous vaccination against diphtheria, tetanus, pertussis, Hemophilus influenzae type b and/or Streptococcus pneumoniae. Locally recommended EPI vaccines to be given at birth are allowed, but should be administered at least one month before the first dose of the study vaccine is administered. Other locally recommended vaccines are allowed, even if concomitantly administered with the study vaccines, but should be documented in the eCRF.

Ages: 6 Weeks to 12 Weeks | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 300 (Actual)
Dates: Start 2011-02-17 (Actual); Primary Completion 2011-07-26 (Actual); Study Completion 2011-07-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Ho Chi Minh City, Vietnam

IPD SHARING:
Plan to Share IPD: Yes
IPD is available via the Clinical Study Data Request site (click on the link provided below)
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: IPD is available via the Clinical Study Data Request site (click on the link provided below)
Access Criteria: Access is provided after a research proposal is submitted and has received approval from the Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an extension can be granted, when justified, for up to another 12 months.
URL: https://clinicalstudydatarequest.com/Posting.aspx?ID=473

REFERENCES:
- [Background] Huu TN, Toan NT, Tuan HM, Viet HL, Le Thanh Binh P, Yu TW, Shafi F, Habib A, Borys D. Safety and reactogenicity of primary vaccination with the 10-valent pneumococcal non-typeable Haemophilus influenzae protein D conjugate vaccine in Vietnamese infants: a randomised, controlled trial. BMC Infect Dis. 2013 Feb 21;13:95. doi: 10.1186/1471-2334-13-95. PMID 23432812
- [Background] Tran NH et al. Safety and reactogenicity of the 10-valent pneumococcal non-typeable Haemophilus influenzae protein D conjugate vaccine (PHiD-CV) co-administered with DTPa-HBV-IPV/Hib in Vietnamese infants. Abstract presented at the ICID, Bangkok, Thailand, June 13-16, 2012.
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Clinical Study Report: 113151 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 113151 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 113151 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 113151 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 113151 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 113151 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 300 subjects were enrolled in this study. 2 subjects among the 101 subjects in the Infanrix Hexa Group were not vaccinated due to consent withdrawal.
Groups:
- Synflorix+Infanrix Hexa Group: Healthy male or female subjects who received the Synflorix™ vaccine, intramuscularly in the right thigh, co-administered along with the Infanrix hexa™ vaccine, intramuscularly in the left thigh, according to a 3-dose schedule at 2, 3 and 4 months of age.
- Infanrix Hexa Group: Healthy male or female subjects who received the Infanrix hexa™ vaccine alone, administered intramuscularly in the left thigh, according to a 3-dose schedule at 2, 3 and 4 months of age.
Period: Overall Study
Arm/Group | Synflorix+Infanrix Hexa Group | Infanrix Hexa Group
Started | 199 | 99
Completed | 193 | 99
Not Completed | 6 | 0
Not completed — Adverse Event | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0
Not completed — Protocol Violation | 2 | 0
Not completed — Lost to Follow-up | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Synflorix+Infanrix Hexa Group | Infanrix Hexa Group | Total
Number analyzed (Participants) | 199 | 99 | 298
Age, Continuous [Mean (Standard Deviation); unit: Weeks] | 8.8 (1.24) | 8.7 (1.11) | 8.77 (1.20)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 93 | 37 | 130
  Male | 106 | 62 | 168

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects With Grade 3 Symptoms (Solicited and Unsolicited)
Description: The incidence and nature of Grade 3 symptoms (solicited and unsolicited) reported during the 31-day post-vaccination period following each dose and across doses are presented.
Time Frame: Within the 31-day (Days 0-30) after each dose and across doses
Population: The analysis was performed on the Total Vaccinated cohort, which included all vaccinated subjects with at least one vaccine administration documented and with the symptom sheet filled in.
Measure: Count of Participants; unit: Participants
Arm/Group | Synflorix+Infanrix Hexa Group | Infanrix Hexa Group
Number analyzed (Participants) | 197 | 99
Participants
  Any symptom Dose 1 | 24 | 3
  Any symptom Dose 2: number analyzed (Participants) | 193 | 99
  Any symptom Dose 2 | 18 | 3
  Any symptom Dose 3: number analyzed (Participants) | 193 | 99
  Any symptom Dose 3 | 6 | 3
  Any symptom Across doses | 32 | 9
  General symptoms Dose 1 | 5 | 1
  General symptoms Dose 2: number analyzed (Participants) | 193 | 99
  General symptoms Dose 2 | 7 | 1
  General symptoms Dose 3: number analyzed (Participants) | 193 | 99
  General symptoms Dose 3 | 1 | 1
  General symptoms Across doses | 10 | 3
  Local symptoms Dose 1 | 23 | 2
  Local symptoms Dose 2: number analyzed (Participants) | 193 | 99
  Local symptoms Dose 2 | 15 | 2
  Local symptoms Dose 3: number analyzed (Participants) | 193 | 99
  Local symptoms Dose 3 | 5 | 2
  Local symptoms Across doses | 28 | 6

2. Secondary Outcome: Number of Subjects Reporting Any and Grade 3 Solicited Local Symptoms
Description: Solicited local symptoms assessed include pain, redness and swelling. Grade 3 pain was defined as crying when limb was moved/spontaneously painful. Grade 3 swelling/redness was defined as swelling/redness larger than (>) 30 millimeters (mm). "Any" is defined as incidence of the specified symptom regardless of intensity.
Time Frame: During the 4-day (Days 0-3) post-vaccination period following each dose
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Synflorix+Infanrix Hexa Group | Infanrix Hexa Group
Number analyzed (Participants) | 197 | 99
Participants
  Any Pain Dose 1 | 116 | 34
  Grade 3 Pain Dose 1 | 22 | 1
  Any Redness Dose 1 | 48 | 13
  Grade 3 Redness Dose 1 | 3 | 0
  Any Swelling Dose 1 | 47 | 10
  Grade 3 Swelling Dose 1 | 3 | 1
  Any Pain Dose 2: number analyzed (Participants) | 193 | 99
  Any Pain Dose 2 | 101 | 31
  Grade 3 Pain Dose 2: number analyzed (Participants) | 193 | 99
  Grade 3 Pain Dose 2 | 12 | 2
  Any Redness Dose 2: number analyzed (Participants) | 193 | 99
  Any Redness Dose 2 | 49 | 19
  Grade 3 Redness Dose 2: number analyzed (Participants) | 193 | 99
  Grade 3 Redness Dose 2 | 1 | 0
  Any Swelling Dose 2: number analyzed (Participants) | 193 | 99
  Any Swelling Dose 2 | 44 | 12
  Grade 3 Swelling Dose 2: number analyzed (Participants) | 193 | 99
  Grade 3 Swelling Dose 2 | 2 | 0
  Any Pain Dose 3: number analyzed (Participants) | 193 | 99
  Any Pain Dose 3 | 68 | 27
  Grade 3 Pain Dose 3: number analyzed (Participants) | 193 | 99
  Grade 3 Pain Dose 3 | 4 | 0
  Any Redness Dose 3: number analyzed (Participants) | 193 | 99
  Any Redness Dose 3 | 38 | 12
  Grade 3 Redness Dose 3: number analyzed (Participants) | 193 | 99
  Grade 3 Redness Dose 3 | 1 | 1
  Any Swelling Dose 3: number analyzed (Participants) | 193 | 99
  Any Swelling Dose 3 | 29 | 12
  Grade 3 Swelling Dose 3: number analyzed (Participants) | 193 | 99
  Grade 3 Swelling Dose 3 | 2 | 1

3. Secondary Outcome: Number of Subjects Reporting Any, Grade 3 and Related Solicited General Symptoms
Description: Solicited general symptoms assessed include drowsiness, fever (defined as axillary temperature ≥ 37.5°C), irritability, and loss of appetite. Grade 3 drowsiness was defined as drowsiness which prevented normal everyday activities. Grade 3 fever was defined as fever (axillary temperature) above (>) 39.5 degree Celsius (°C). Grade 3 irritability was defined as crying that could not be comforted/preventing normal activity. Grade 3 loss of appetite was defined as the subject not eating at all. "Any" is defined as incidence of the specified symptom regardless of intensity or relationship to study vaccination.
Time Frame: During the 4-day (Days 0-3) post-vaccination period following each dose
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Synflorix+Infanrix Hexa Group | Infanrix Hexa Group
Number analyzed (Participants) | 197 | 99
Participants
  Any Drowsiness Dose 1 | 75 | 19
  Grade 3 Drowsiness Dose 1 | 3 | 0
  Related Drowsiness Dose 1 | 60 | 15
  Any Fever Dose 1 | 147 | 36
  Grade 3 Fever Dose 1 | 0 | 0
  Related Fever Dose 1 | 142 | 34
  Any Irritability Dose 1 | 155 | 53
  Grade 3 Irritability Dose 1 | 4 | 1
  Related Irritability Dose 1 | 146 | 51
  Any Loss of appetite Dose 1 | 109 | 40
  Grade 3 Loss of appetite Dose 1 | 0 | 0
  Related Loss of appetite Dose 1 | 86 | 31
  Any Drowsiness Dose 2: number analyzed (Participants) | 193 | 99
  Any Drowsiness Dose 2 | 53 | 10
  Grade 3 Drowsiness Dose 2: number analyzed (Participants) | 193 | 99
  Grade 3 Drowsiness Dose 2 | 0 | 0
  Related Drowsiness Dose 2: number analyzed (Participants) | 193 | 99
  Related Drowsiness Dose 2 | 52 | 8
  Any Fever Dose 2: number analyzed (Participants) | 193 | 99
  Any Fever Dose 2 | 108 | 16
  Grade 3 Fever Dose 2: number analyzed (Participants) | 193 | 99
  Grade 3 Fever Dose 2 | 0 | 0
  Related Fever Dose 2: number analyzed (Participants) | 193 | 99
  Related Fever Dose 2 | 105 | 15
  Any Irritability Dose 2: number analyzed (Participants) | 193 | 99
  Any Irritability Dose 2 | 112 | 36
  Grade 3 Irritability Dose 2: number analyzed (Participants) | 193 | 99
  Grade 3 Irritability Dose 2 | 6 | 0
  Related Irritability Dose 2: number analyzed (Participants) | 193 | 99
  Related Irritability Dose 2 | 110 | 32
  Any Loss of appetite Dose 2: number analyzed (Participants) | 193 | 99
  Any Loss of appetite Dose 2 | 94 | 25
  Grade 3 Loss of appetite Dose 2: number analyzed (Participants) | 193 | 99
  Grade 3 Loss of appetite Dose 2 | 0 | 0
  Related Loss of appetite Dose 2: number analyzed (Participants) | 193 | 99
  Related Loss of appetite Dose 2 | 90 | 23
  Any Drowsiness Dose 3: number analyzed (Participants) | 193 | 99
  Any Drowsiness Dose 3 | 25 | 5
  Grade 3 Drowsiness Dose 3: number analyzed (Participants) | 193 | 99
  Grade 3 Drowsiness Dose 3 | 0 | 0
  Related Drowsiness Dose 3: number analyzed (Participants) | 193 | 99
  Related Drowsiness Dose 3 | 21 | 4
  Any Fever Dose 3: number analyzed (Participants) | 193 | 99
  Any Fever Dose 3 | 63 | 12
  Grade 3 Fever Dose 3: number analyzed (Participants) | 193 | 99
  Grade 3 Fever Dose 3 | 0 | 1
  Related Fever Dose 3: number analyzed (Participants) | 193 | 99
  Related Fever Dose 3 | 60 | 12
  Any Irritability Dose 3: number analyzed (Participants) | 193 | 99
  Any Irritability Dose 3 | 71 | 31
  Grade 3 Irritability Dose 3: number analyzed (Participants) | 193 | 99
  Grade 3 Irritability Dose 3 | 1 | 0
  Related Irritability Dose 3: number analyzed (Participants) | 193 | 99
  Related Irritability Dose 3 | 69 | 29
  Any Loss of appetite Dose 3: number analyzed (Participants) | 193 | 99
  Any Loss of appetite Dose 3 | 67 | 21
  Grade 3 Loss of appetite Dose 3: number analyzed (Participants) | 193 | 99
  Grade 3 Loss of appetite Dose 3 | 0 | 0
  Related Loss of appetite Dose 3: number analyzed (Participants) | 193 | 99
  Related Loss of appetite Dose 3 | 60 | 19

4. Secondary Outcome: Number of Subjects With Unsolicited Adverse Events (AEs)
Description: An unsolicited AE is any untoward medical occurrence in a clinical investigation subject, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. "Any" is defined an incidence of an unsolicited AE regardless of intensity or relationship to study vaccination.
Time Frame: During the 31-day (Days 0-30) follow-up period after each dose
Population: The analysis was performed on the Total Vaccinated cohort, which included all vaccinated subjects with at least one vaccine administration documented.
Measure: Count of Participants; unit: Participants
Arm/Group | Synflorix+Infanrix Hexa Group | Infanrix Hexa Group
Number analyzed (Participants) | 199 | 99
Participants | 57 | 37

5. Secondary Outcome: Number of Subjects With Serious Adverse Events (SAEs)
Description: SAEs assessed include medical occurrences that result in death, are life-threatening, require hospitalization or prolongation of hospitalization or result in disability/incapacity.
Time Frame: After the first vaccination up to study end (From Month 0 to Month 3)
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | Synflorix+Infanrix Hexa Group | Infanrix Hexa Group
Number analyzed (Participants) | 199 | 99
Participants | 9 | 6

ADVERSE EVENTS:
Time Frame: Solicited local and general symptoms: during the 4-day (Day 0 - Day 3) post-vaccination period; Unsolicited AEs: during the 31-day (Day 0 - Day 30) post-vaccination period; SAEs: after the first vaccination up to study end (from Month 0 to Month 3).
Arm/Group | Synflorix+Infanrix Hexa Group | Infanrix Hexa Group
Serious Adverse Events (participants affected / at risk) | 9/199 | 6/99
Other Adverse Events (participants affected / at risk) | 195/199 | 91/99
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Synflorix+Infanrix Hexa Group (N=199) | Infanrix Hexa Group (N=99)
Kawasaki's disease (Vascular disorders) | 1 | 0
Autoimmune thrombocytopenia (Blood and lymphatic system disorders) | 1 | 0
Coagulopathy (Blood and lymphatic system disorders) | 1 | 0
Convulsion (Nervous system disorders) | 1 | 0
Febrile convulsion (Nervous system disorders) | 1 | 0
Hydronephrosis (Renal and urinary disorders) | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 2
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 | 1
Bronchiolitis (Infections and infestations) | 2 | 3
Superinfection fungal (Infections and infestations) | 1 | 2
Diarrhoea infectious (Infections and infestations) | 1 | 0
Oral candidiasis (Infections and infestations) | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 1 | 0
Urinary tract infection (Infections and infestations) | 0 | 1
Viral infection (Infections and infestations) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs:
Term (organ system) | Synflorix+Infanrix Hexa Group (N=199) | Infanrix Hexa Group (N=99)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 | 5
Pain (General disorders) | 137/197 | 45
Redness (General disorders) | 90/197 | 29
Swelling (General disorders) | 80/197 | 21
Drowsiness (General disorders) | 95/197 | 26
Fever (Axillary) (General disorders) | 172/197 | 50
Irritability (General disorders) | 169 | 63
Loss of appetite (General disorders) | 141/197 | 50
Upper respiratory tract infection (Infections and infestations) | 20 | 8
Bronchiolitis (Infections and infestations) | 9 | 9

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.